CLINICAL TRIAL: NCT07013370
Title: Immunoglobulin-specific Prophylaxis Against Citomegalovirus Infections in Immunocompromised Children Undergoing Allogeneic Hematopoietic Stem Cell Transplantation
Brief Title: Immunoglobiulin-specific Prophylaxis of Citomegalovirus Infections in Immunocompromised Children Undergoing Allogeneic Hematopoietic Stem Cell Transplantation
Status: Recruiting | Type: Observational
Sponsor: Antonello Di Paolo, M.D., Ph.D. (Other)
Collaborators: IRCCS Burlo Garofolo (Other)
Responsible Party: Sponsor-Investigator, Antonello Di Paolo, M.D., Ph.D., Assistant Professor of Pharmacology, University of Pisa
Organization: University of Pisa (Other)
Other Study IDs: 1105/2015_BG
Record Dates: First submitted 2025-06-02; First posted 2025-06-10 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-06

CONDITIONS: Immunoglobulin Prophylaxis; Cytomegalovirus Infections; Allogeneic Hematopoietic Stem Cell Transplantation; Transplant-Related Disorder
Keywords: Cytomegalovirus; allo-HSCT; Transplant-Related mortality
MeSH Terms: conditions — Cytomegalovirus Infections

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Control Group: Pediatric allo-HSCT recipients who have not received CMV-specific immunoglobulin prophylaxis after transplantation.
- Immunoprophylaxis Group: Pediatric allo-HSCT recipients who received an anti-CMV prophylaxis with immunoglobulin (Megalotect)
  Interventions: Biological: Anti-CMV immunoglobulins [Megalotect (R)]

INTERVENTIONS:
Biological: Anti-CMV immunoglobulins [Megalotect (R)] — Children received an anti-CMV immunoglobulin to prevent viral infections
  Groups: Immunoprophylaxis Group

SUMMARY:
Human cytomegalovirus (CMV) is a globally prevalent, human-specific herpesvirus characterised by a lifelong latency after primary infection, an often asymptomatic reactivation and affecting up to 100% of adults based on region and age. CMV reactivation has serious risks for immunocompromised patients, especially those undergoing allogeneic hematopoietic stem cell transplantation (HSCT). In these patients, CMV can lead to graft failure, multiorgan disease, increased risk of other infections, GVHD, post-transplant lymphoproliferative disorders, and higher transplant-related mortality (TRM). Although antiviral prophylaxis, CMV infection occurs in 38-80% of HSCT recipients, but current antiviral drugs are insufficiently effective and they are associated with adverse effects. Furthermore, treatment failure is due to the high genetic variability of CMV. The protective role of virus-specific antibodies remains under debate. Some studies suggest that high neutralizing antibody titers protect transplant recipients from CMV, while others highlight the importance of T-cell responses. However, recent animal studies showed that humoral immunity alone can prevent CMV reactivation, even without T or NK cells. In solid-organ transplant patients, antibody titers ≥480 have been linked to reduced infection, shorter treatment, and full protection from CMV disease. Although the use of anti-CMV immunoglobulin remains controversial, the IRCCS Burlo Garofolo has used it as post-transplant prophylaxis and second-line treatment for over a decade.

The main objective of their study was to assess whether CMV-specific immunoglobulin prophylaxis reduces CMV incidence and severity in pediatric HSCT patients. Secondary goals included evaluating its effect on transplant outcomes and its efficacy across different ethnic groups. A population pharmacokinetic (POP/PK) study was also conducted to better understand the drug's distribution and elimination and to identify factors influencing its pharmacokinetics in patients.

DETAILED DESCRIPTION:
The study will enroll all patients who received standard myeloablative conditioning. GVHD prophylaxis consisting of tacrolimus and, for unrelated donors, rabbit ATG and mycophenolate mofetil. Haploidentical transplants initially used in vivo T-cell depletion with post-transplant cyclophosphamide, later replaced by ex vivo αβ+/CD19+ T-cell depletion.

Outcomes included overall survival (OS), relapse-related mortality (RRM), and GVHD, defined by standard grading systems. Immune reconstitution was measured by CD4+ T-lymphocyte counts, with ≥500 cells/μL in two readings within 100 days post-HSCT considered adequate. Follow-up continued until death or last contact, with a minimum duration of 12 months for survivors.

Viral Load Detection

CMV DNAemia was quantified in whole blood using real-time PCR (CMV ELITe MGB Kit). Monitoring occurred twice weekly during hospitalization, then weekly in outpatient visits until immune reconstitution and end of immunosuppression.

CMV-Specific Immunoglobulin Prophylaxis and Treatment

Prophylaxis was administered using Cytomegatect® (Biotest Pharma GmbH), beginning on day 3 of conditioning and continued biweekly during hospitalization. Post-discharge, it was given at each hospital admission until CD4+ normalization. If DNAemia appeared, a 3-5 day "boost" treatment was given based on risk assessment. Non-responders (based on viral load behavior) discontinued treatment. In cases of CMV disease, dosing and treatment duration were tailored. Cytomegatect was dosed by weight: 1000 U (<10 kg), 2000 U (10-25 kg), 3000 U (25-50 kg), and 4000 U (>50 kg).

Foscarnet was used as first-line therapy within the first post-transplant month. Ganciclovir or valganciclovir was introduced after engraftment. Second-line options included cidofovir, letermovir, and maribavir. Advanced therapies involved NK or CD45RO+ lymphocyte infusions. CMV IgG levels were monitored 24-72 hours after each infusion for inpatients and before administration for outpatients.

CMV-Related Complications

CMV-related complications were classified per Ljungman et al.'s updated definitions. CMV infection referred to virus detection in body fluids or tissues. DNAemia denoted CMV DNA presence in blood. Primary infection was the first detection in previously unexposed patients; recurrent infections occurred after a 4-week CMV-negative interval. Refractory infections showed persistent or increasing viral load despite at least two weeks of treatment. CMV disease followed existing consensus criteria.

Statistical and POP/PK Analyses

Continuous variables were summarized by means or medians with interquartile ranges, depending on distribution (tested via Shapiro-Wilk). Categorical variables were presented as counts and percentages. Group comparisons were performed using chi-square tests for qualitative variables and Wilcoxon tests for continuous ones. Kaplan-Meier curves and log-rank tests assessed survival outcomes. Differences in pharmacokinetics between occasions were evaluated with ANOVA.

Plasma concentrations of anti-CMV immunoglobulin were analyzed using a nonlinear mixed-effects modeling approach via Monolix 2023.1. Mono-, bi-, and tri-compartmental models with various error structures were evaluated. Covariates (age, weight, creatinine clearance) were assessed for influence on model performance, which was judged based on objective function value (OFV), standard errors, and residual distributions. Individual elimination half-lives were calculated as t½ = (0.693 × Vi) / Cli, where Vi and Cli are individual volume of distribution and clearance values

ELIGIBILITY:
Inclusion Criteria:

* Children who underwent allogeneic HSCT due to any condition

Exclusion Criteria:

* Positive personal records of immunoglobulin-related adverse reactions
* CMV reactivation before the CMV-specific immunoglobulin prophylaxis onset
* adoptive cellular post-HSCT immunotherapy for any indication

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children who underwent allogeneic HSCT due to any condition
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2025-06-02 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-06-02 (Estimated)

PRIMARY OUTCOMES:
CMV reactivation and infection | 12 months since allo-HSCT
  The rate of viral reactivation and infection in children undergoing all-HSCT

SECONDARY OUTCOMES:
Overall Survival | 12 months since allo-HSCT
  The rate of overall survival since allo-HSCT
Hospital stay | 12 months since allo-HSCT
  The lenght of hospital stay after allo-HSCT
Immunological recovery | 12 months since allo-HSCT
  The percentage of patients in who the function of CD4+ lymphocytes was restored
GVHD incidence | 12 months since allo-HSCT
  The percentage of patients who experienced a GVHD

CONTACTS AND LOCATIONS:
Overall Officials: Natalia Maximova, MD, Principal Investigator — IRCCS Burlo Garofolo - Trieste - ITALY
Locations (1):
- IRCCS Burlo Garofolo, Trieste, Italy

IPD SHARING:
Plan to Share IPD: Undecided
Data sharing will be discussed case by case upon reasonable request and after local IRB approval.